CLINICAL TRIAL: NCT03739541
Title: A Phase I, Open-label, Study of the Absorption, Metabolism and Excretion, of [14C]-Benznidazole (BNZ) Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Benznidazole Absorption, Metabolism and Excretion Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exeltis France (Unknown)
Collaborators: Insud Pharma (Industry)
Responsible Party: Sponsor
Organization: Insud Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LPRI747-103
Record Dates: First submitted 2018-07-06; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-09

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]-Benznidazole (Experimental): A single dose of 100 mg [14C]-BNZ, orally administered on Day 1 following an overnight fast.
  Interventions: Drug: [14C]-Benznidazole

INTERVENTIONS:
Drug: [14C]-Benznidazole — A single dose level of 100 mg; 200 μCi (7.4 MBq)
  Other Names: BNZ

SUMMARY:
This Phase I ADME study will be conducted to evaluate the pharmacokinetics of benznidazole.

DETAILED DESCRIPTION:
This will be a single-site, open-label, non-randomized, single oral dose absorption, metabolism and excretion study in healthy male subjects. Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to dosing on Day 1. Subjects will be admitted into the Clinical Research Unit (CRU) on Day -1. Subjects will be confined to the CRU until at least Day 11 (240 hours postdose), and will be discharged from the CRU on Day 11 if all the following discharge criteria are met: >90% mass balance recovery; OR plasma/blood radioactivity levels below the limit of quantitation for 2 consecutive collections; and <1% of the total radioactive dose recovered in combined excreta (urine and faeces) in 2 consecutive 24-hour periods. If these criteria are not met by Day 11, subjects will remain in the CRU until all discharge criteria are met up to a maximum of Day 15 to continue 24-hour blood, urine and faeces collections for the analysis of total radioactivity, unless otherwise agreed upon by the Sponsor and Investigator. If the discharge criteria are not met by Day 15, subjects may be asked to collect 24-hour excreta samples on up to 2 further occasions on a nonresidential basis to allow extrapolation of urinary and faecal excretion. If needed, the 2 additional 24-hour nonresidential collections will occur on Day 21 (±1 day) and Day 28 (±1 day). If on the second occasion the subject has still not met the desired criterion, then the subject will be discharged from the study, per Investigator and Sponsor decision. Pharmacokinetic samples and radioanalytical samples will be obtained through at least 240 hours postdose, and possibly up to 4 weeks postdose (radioanalytical samples only), in case of not meeting discharge criteria. Samples for metabolite profiling/identification will be obtained through 240 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

1. Males of any race, between 35 and 65 years of age, inclusive, at screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable) at screening or check-in as assessed by the Investigator (or designee).
4. Will agree to use contraception as detailed in Section 7.6.
5. History of a minimum of 1 bowel movement per day.
6. Able to comprehend and willing to sign an Inform Consent Form and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. History of dermatological conditions within the 6 months prior to dosing, such as rash, pruritus, and dermatitis, as determined by the Investigator (or designee).
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). Cholecystectomy is acceptable.
5. History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
6. Alcohol consumption of >28 units per week for males. One unit of alcohol equals

   ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
7. Positive alcohol breath test or positive urine cotinine test result, or positive urine drug screen (confirmed by repeat) at screening or check-in.
8. Positive hepatitis panel and/or positive human immunodeficiency virus test (Appendix 3).
9. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to check-in.
10. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to check-in, unless deemed acceptable per Investigator (or designee) and Sponsor decision.
11. Use or intend to use any prescription medications/products within 14 days prior to check-in, unless deemed acceptable by the Investigator (or designee).
12. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the Investigator (or designee).
13. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check-in, unless deemed acceptable per Investigator (or designee) and Sponsor decision.
14. Use of tobacco- or nicotine-containing products within 3 months prior to check-in.
15. Receipt of blood products within 2 months prior to check-in.
16. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
17. Poor peripheral venous access.
18. Have previously completed or withdrawn from this study or any other study investigating BNZ, and have previously received the investigational product.
19. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
20. Subjects who have participated in any clinical trial involving a radiolabelled investigational product within 12 months prior to check-in.
21. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Cmax of BNZ in plasma | Days 1-29
  maximum observed concentration (Cmax) in plasma
Mass balance of [14C]-BNZ | Days 1-29
  Mass balance of [14C]-BNZ in urine and faeces
Chemical structure of [14C]-BNZ metabolites | Days 1-29
  Characterization of the chemical structure and identification of metabolites of [14C]-BNZ in plasma, urine, and faeces
tmax of BNZ in plasma | Days 1-29
  time to maximum concentration (tmax) in plasma
AUC0-t of BNZ in plasma | Days 1-29
  area under the concentration-time curve (AUC) from hour zero to the last measurable concentration (AUC0-t) in plasma
AUC0-∞ of BNZ in plasma | Days 1-29
  AUC from time zero to infinity (AUC0-∞) in plasma
% AUC extrap of BNZ in plasma | Days 1-29
  percentage extrapolation (% AUCextrap) in plasma
t1/2 of BNZ in plasma | Days 1-29
  apparent terminal elimination half-life (t1/2) in plasma
CL/Fof BNZ in plasma | Days 1-29
  apparent oral clearance (CL/F) in plasma
Vz/F of BNZ in plasma | Days 1-29
  volume of distribution during the elimination phase for BNZ (Vz/F) in plasma
Cmax of [14C]-BNZ in plasma | Days 1-29
  maximum observed concentration (Cmax) in plasma
tmax of [14C]-BNZ in plasma | Days 1-29
  time to maximum concentration (tmax) in plasma
AUC0-t of [14C]-BNZ in plasma | Days 1-29
  area under the concentration-time curve (AUC) from hour zero to the last measurable concentration (AUC0-t) in plasma
AUC0-∞ of [14C]-BNZ in plasma | Days 1-29
  AUC from time zero to infinity (AUC0-∞) in plasma
% AUC extrap of [14C]-BNZ in plasma | Days 1-29
  percentage extrapolation (% AUCextrap) in plasma
t1/2 of [14C]-BNZ in plasma | Days 1-29
  apparent terminal elimination half-life (t1/2) in plasma
Cmax of [14C]-BNZ in whole blood | Days 1-29
  maximum observed concentration (Cmax) in whole blood
tmax of [14C]-BNZ in whole blood | Days 1-29
  time to maximum concentration (tmax) in whole blood
AUC0-t of [14C]-BNZ in whole blood | Days 1-29
  area under the concentration-time curve (AUC) from hour zero to the last measurable concentration (AUC0-t) in whole blood
AUC0-∞ of [14C]-BNZ in whole blood | Days 1-29
  AUC from time zero to infinity (AUC0-∞) in whole blood
% AUCextrap of [14C]-BNZ in whole blood | Days 1-29
  percentage extrapolation (% AUCextrap) in whole blood
t1/2 of [14C]-BNZ in whole blood | Days 1-29
  apparent terminal elimination half-life (t1/2) in whole blood
Total radioactivity AUC ratio | Days 1-29
  Total radioactivity AUC ratio (blood/plasma)

SECONDARY OUTCOMES:
The incidence and severity of Adverse Events (AEs) | Days 1-29
  The incidence of AEs will be presented by severity and by association with the study drug as determined by the Investigator (or designee).
The incidence of laboratory abnormalities (haematology) | Days 1-29
  The incidence of laboratory abnormalities will be measured based on haematology test result.
The incidence of laboratory abnormalities (clinical chemistry) | Days 1-29
  The incidence of laboratory abnormalities will be measured based on clinical chemistry test result.
The incidence of laboratory abnormalities (urinalysis) | Days 1-29
  The incidence of laboratory abnormalities will be measured based on urinalysis test result.
Measurement of QT interval (QTcB) | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); QT interval calculated using the Bazett correction (QTcB) in millisecond
Measurement of QT interval (QTcF) | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); QT interval calculated using the Fridericia correction (QTcF) in millisecond
Measurement of PR intervals | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); PR intervals in millisecond.
Measurement of QT intervals | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); QT intervals in millisecond
Measurement of QRS duration | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); QRS duration in millisecond
Measurement of RR | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); RR in millisecond
Measurement of heart rate | Days 1-29
  Measure of 12-lead electrocardiogram (ECG); heart rate in beats per minute (BPM)
Measurement of blood pressure | Days 1-29
  Measure of supine systolic and diastolic blood pressure ( both in mmHg)
Measurement of Physical Examination | Days 1-29
  Weight (in kilograms) and Height (in centimeters) will be measured
Measurement of supine pulse rate | Days 1-29
  supine pulse rate (in beats/minute)
Measurement body temperature | Days 1-29
  oral body temperature (in Degree Celsius)
Measurement of Weight | Days 1-29
  weight (in kilograms)
Measurement of Height | Days 1-29
  height (in centimeters) w

CONTACTS AND LOCATIONS:
Overall Officials: Sunu Valasseri, MBBS, MSc, Principal Investigator — Covance
Locations (1):
- Covance, Leeds, United Kingdom